CLINICAL TRIAL: NCT06344546
Title: Metabolic Pathway Analysis in Refeeding Syndrome: a Nested Explorative Metabolomics Substudy of the GUTPHOS Multicenter Observational Study (GUTPHOS-Metabolomics)
Brief Title: Metabolic Pathway Analysis in Intensive Care Unit Patients With Refeeding Syndrome
Status: Completed | Type: Observational
Sponsor: Karolinska University Hospital (Other)
Collaborators: Foggia Hospital (Unknown); Faculty Hospital Kralovske Vinohrady (Other Government)
Responsible Party: Principal Investigator, Martin Sundstrom Rehal, Principal Investigator, Karolinska University Hospital
Other Study IDs: K 2023-10247
Record Dates: First submitted 2024-03-07; First posted 2024-04-03 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Critical Illness; Refeeding Syndrome; Hypophosphatemia
MeSH Terms: conditions — Critical Illness; Refeeding Syndrome; Hypophosphatemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples (2 ml daily for first 7 days in ICU).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Refeeding hypophosphatemia: ICU patients who fulfill diagnostic criteria for refeeding hypophosphatemia.
  Interventions: Diagnostic Test: Metabolomics
- Controls: ICU patients without refeeding hypophosphatemia. Controls selected to match for sex, age, severity of illness and nutritional delivery prior to refeeding hypophosphatemia.
  Interventions: Diagnostic Test: Metabolomics

INTERVENTIONS:
Diagnostic Test: Metabolomics — Analysis of the metabolome in plasma samples.

SUMMARY:
The overall aim of the study is to improve understanding of refeeding syndrome (RFS) in patients admitted to the intensive care unit (ICU) using metabolomics. Patients are included as part of a prospective multicenter observational study on phosphate disorders in the ICU. Blood samples are collected day 1-7 of ICU stay. Samples from patients who develop refeeding hypophosphatemia and matched controls without hypophosphatemia are analysed for metabolomics and proteomics. Untargeted analyses will be performed to identify the affected metabolic pathways. The investigators will also perform AUROC analyses to identify potential biomarkers for early detection of RFS.

DETAILED DESCRIPTION:
A nested case-control study situated within GUTPHOS Part B: A prospective, multicenter non-interventional cohort study investigating the incidence of abnormal phosphate levels and associated outcomes in adult patients admitted to the ICUs of participating sites. Inclusion/exclusion criteria for GUTPHOS Part B are described in the separate study protocol.

At sites participating in the nested substudy, an additional 2 ml EDTA blood sample is drawn once daily in all patients included in GUTPHOS Part B from ICU admission up to a maximum of calendar day 7 in ICU. The sampling for metabolomics analysis should be performed in close proximity with daily routine blood tests, and always before treatment of hypophosphatemia with phosphate supplementation or restricted nutritional intake. Plasma samples are obtained through centrifugation within 20 minutes and frozen to -80 degrees Celcius within 60 minutes until analysis. The timing and handling of samples according to standard operating procedures will be documented on a separate case report form.

In ICU patients diagnosed with refeeding hypophosphatemia, comprehensive metabolomic profiling is performed in the plasma sample from ICU admission and the sample drawn in conjunction to the blood phosphate measurement diagnostic of RH.

Cases with RH are matched in a 1:1 ratio to ICU patients without RH. Controls are matched according to sex, age, illness severity on admission and energy delivery (kcal/kg adjusted body weight) in the 24 hours preceding the diagnosis of RH.

Refeeding hypophosphatemia is defined as new onset hypophosphatemia (<0.65 mmol/L) within 72 hours from the start of medical nutrition therapy, with a drop of >0.16 mmol/L from any previous Pi value during ICU stay and where no other likely cause of hypophosphatemia is present.

ELIGIBILITY:
Inclusion Criteria:

* Admission to ICU during the study period
* Age ≥18 years

Exclusion Criteria:

* Age <18 years
* Patients with restrictions of care such as "no intubation" or "no renal replacement therapy" on ICU admission and patients admitted for treatment as organ donors
* Continuous chronic home ventilation for neuromuscular disease;
* Declined participation or informed consent (if the local ethics committee requests the latter for this non-interventional study);
* Readmission to ICU during the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the intensive care unit.
Sampling Method: Non-Probability Sample
Enrollment: 218 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-06-02 (Actual); Study Completion 2024-06-02 (Actual)

PRIMARY OUTCOMES:
Metabolomics | Onset of RFS, within the first 7 days in ICU.
  The plasma metabolome (>300 metabolites related to cell metabolism) will be characterized by mass spectroscopy from blood samples taken at the onset of refeeding syndrome (RFS) and analyzed for specific alterations in metabolic pathways associated with RFS in an untargeted approach.

SECONDARY OUTCOMES:
Metabolomics | Prior to onset of RFS, within the first 7 days in ICU.
  Potential biomarkers in the plasma metabolome (>300 metabolites related to cell metabolism) associated with the development of refeeding syndrome (RFS) will be identified through principal component analysis and ROC curve analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Olav Rooyackers, PhD, Study Chair — Karolinska University Hospital
Locations (4):
- University Hospital Královské Vinohrady, Prague, Czechia
- University Hospital Policlinico of Foggia, Foggia, Italy
- Sweden (2):
  - Karolinska University Hospital, Huddinge, Stockholm County
  - Karolinska Universitetssjukhuset Solna, Stockholm

IPD SHARING:
Plan to Share IPD: Undecided